CLINICAL TRIAL: NCT02278406
Title: Employing Near Infrared Spectroscopy to Non-invasively Assess Changes in Cerebral Perfusion in Response to Subthalamic Deep Brain Stimulation
Brief Title: Non-invasive Measurement of Brain Oxygen Levels in People With Subthalamic Deep Brain Stimulators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Ron Alterman, Professor of Neurosurgery, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2013P000117
Record Dates: First submitted 2014-10-28; First posted 2014-10-30 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Deep brain stimulator; dbs
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Parkinson's patients with DBS (Experimental): Patients with Parkinson's Disease who are at least 3-months post subthalamic deep brain stimulator surgery
  Interventions: Other: Deep brain stimulator

INTERVENTIONS:
Other: Deep brain stimulator — We will measure brain oxygen levels with a non-invasive near infrared spectroscopy device.

SUMMARY:
The purpose of this study is to determine if deep brain stimulation can change brain oxygen levels in people with Parkinson's Disease. Measurements will be taken using a non-invasive device while subjects are both on and off their medications, and while their stimulator is in the on and off setting.

DETAILED DESCRIPTION:
The investigators will study the effects of electrical stimulation at the subthalamic nucleus on frontal cerebral perfusion in 10 patients with advanced PD who have already undergone successful STN DBS (Medtronic, Inc., Minneapolis, MN) surgery as evidenced by a 20% or greater improvement in their Unified Parkinson's disease rating scale (UPDRS) motor sub-score (UPDRS-III) with stimulation on vs off, three or more months after surgery. The UPDRS-III is a widely employed and validated rating scale of Parkinson's disease symptom severity that is based on the neurological examination. For the purposes of this study, a movement disorders neurologist will perform all of the neurological assessments. Patients must also be demonstrated to be cognitively intact as evidenced by a Montreal Cognitive Assessment (MoCA) Score of 24 or greater.

This is an experimental study in which we will compare frontal cerebral perfusion (measured non-invasively with the NIRS device) and UPDRS-III scores (as determined by neurological examination) in four clinical states: medications off/stimulation off; medication off/stimulation on; medication on/stimulation off; and medications on/stimulation on.

The primary question to be answered is: Can we detect significant changes in cerebral perfusion with the NIRS device in response to subthalamic stimulation delivered via implanted DBS devices?

This pilot study will be conducted in 10 PD patients who have undergone successful DBS surgery in the past. The study will be completed in one day as detailed below and will take about 6 hours to complete.

Patients will arrive to the movement disorders center on the morning of their scheduled study visit having discontinued their medications from the night before (12 hours 'off"). They will arrive with their stimulators on and set to the therapeutic parameters. Dr. Shih will perform a neurological examination and determine the UPDRS-III score in this, the off med/on stim state.

In order to perform the NIRS/perfusion measurements the subject will be fitted with a multipart plastic helmet, which holds a number of optical fibers against the surface of the subject's head. This helmet will be adjusted to fit comfortably. Additional probes will be positioned on the fingers in order to monitor peripheral blood oxygenation (i.e. pulse oximetry) to ensure that any changes observed in cerebral perfusion are due to changes in brain physiology, not a general physiological factor. The fibers are connected to 32 low power infrared laser diodes. The power emitted by these lasers is far below the typical maximum permissible exposure (MPE) level for skin exposure to a laser beam, as indicated by the American National Standards Institute, and subjects will not feel any effect from them. The laser light will be pointed at the top of their head, and there will be no risk to their eyes. The initial cerebral perfusion measurement will be made.

The patient's DBS devices will then be turned off and 60 min will be allowed to pass, allowing for washout of both the clinical and CBF effects of DBS. During this time, cerebral oxygenation will be monitored and documented every five minutes. At the end of this period the UPDRS-III score will be determined (off meds/off stim) and recorded, confirming a washout of the clinical effects. The DBS will then be turned on employing the settings employed for therapy except that the stimulation frequency will be set to 20Hz, a low frequency that is known not to be therapeutically effective in PD. All other settings will be maintained constant. Again, the cerebral oxygenation will be recorded every 5 min for 60 min after which the UPDRS-III score will be recorded The DBS will then be reprogrammed to the patient's steady state therapeutic settings, the cerebral oxygenation will be recorded every 5 min for 60 min, and at the end of the 60 min period the UPDRS-III score will be recorded again, completing the on stimulation/off medication evaluation. The patient will then be instructed to take his/her usual dose of medications, and will be sent for lunch for one hour. After lunch, the patient will return in the on medication/on stimulation state, the NIRS and pulse oximetry probes will be reapplied, and the process described for the off medication state will be repeated in the on medication state. After the on medication assessments are completed the patient will be sent home with his/her devices on and set to their therapeutic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* Diagnosis of Idiopathic Parkinson's disease made by a movement disorders neurologist.
* At least 3 months status-post bilateral subthalamic deep brain stimulation surgery
* Positive response to STN DBS as evidenced by >20% improvement in UPDRS-III score after surgery as determined by a movement disorders neurologist.
* Cognitively intact as demonstrated with a MOCA > 24.
* Signed informed consent.

Exclusion Criteria:

* Failure to meet all of the inclusion criteria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Brain oxygen levels | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States